CLINICAL TRIAL: NCT06744842
Title: Investigation of the Effect of Ultrasound-Guided Genicular Nerve Block on Knee Joint Proprioception in Patients with Chronic Knee Osteoarthritis
Brief Title: Effect of Genicular Nerve Block on Proprioception in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Handan Elif Nur BAYRAKTAR, specialist, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANKARA-PMR-BEYZA-01
Record Dates: First submitted 2024-11-24; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis
Keywords: Genicular nerve block; Proprioception; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genicular Nerve Block Group (Experimental): A nerve block will be performed on 22 patients using lidocaine injection under ultrasound guidance. After obtaining informed consent, the procedure will be carried out following sterilization, with 2% lidocaine hydrochloride injected at a total volume of 6 mL, distributed as 2 mL for each of the superomedial, superolateral, and inferomedial branches of the genicular nerve. After the injection, bleeding control will be performed, and the procedure will be concluded. All ultrasound-guided injections will be performed by a single physician, and the examination, investigations, treatment, and clinical evaluations of the patients will be conducted by the physicians participating in the study.
  Interventions: Other: genicular nerve block; Other: Exercise
- Exercise group (Active Comparator): Exercise group:
  A home exercise program will be provided, including isometric strengthening exercises for the quadriceps muscles and stretching exercises for the hamstring muscles.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: genicular nerve block — genicular nerve block
  Arms: Genicular Nerve Block Group
Other: Exercise — isometric exercise

SUMMARY:
The study was conducted to investigate the effect of genicular nerve block on pain, quality of life, and proprioception, which are already diminished due to the impact of osteoarthritis in individuals with knee osteoarthritis.

Does genicular nerve block reduce pain and improve the quality of life in patients with knee osteoarthritis? Does genicular nerve block affect proprioception in patients with knee osteoarthritis?

DETAILED DESCRIPTION:
Osteoarthritis (OA) is described as a degenerative joint disease characterized by cartilage erosion, osteophytes, subchondral sclerosis, and changes in the joint capsule, commonly observed in the elderly. Knee osteoarthritis is identified as the most prevalent form, with an increasing prevalence attributed to aging. It is recognized as a leading cause of disability, resulting in reduced quality of life and increased healthcare costs. Major risk factors include age, genetics, obesity, and muscle weakness. Current treatments focus on symptom management, with options including medication, physical therapy, and surgery.

Genicular nerve block is a minimally invasive procedure used to manage knee osteoarthritis pain by administering local anesthetics and corticosteroids near specific genicular nerves under ultrasound guidance. Temporary pain relief for up to three months has been reported, and the procedure is considered well-tolerated.

Proprioception is defined as the sense of joint and limb position, mediated by receptors located in muscles, tendons, and joints. Assessment can be performed through simple methods, such as evaluating the ability to recognize specific joint angles or positions during passive or active movement. Proprioceptive deficits are frequently observed in osteoarthritis, and a better understanding of these changes is suggested to guide treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral primary knee osteoarthritis according to ACR (American College of Rheumatology) criteria.
* Age between 55 and 75 years.
* Presence of knee osteoarthritis classified as Grade 2 or Grade 3 according to the Kellgren-Lawrence grading system on radiographs taken within the last year.
* Knee pain lasting longer than 6 months.
* Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score, total score 48-96

Exclusion Criteria:

* Severe knee trauma within the last 6 months.
* History of surgical operation on the knee region.
* Intra-articular steroid and/or hyaluronate injection into the knee joint within the last 6 months.
* Physical therapy targeting the knee within the last 6 months.
* Regular use of NSAIDs within the last 6 months.
* Presence of acute synovitis.
* Neurological deficits in the lower extremity.
* Presence of an inflammatory disease.
* Poor general health condition (e.g., heart failure, advanced asthma, history of malignancy).
* Any endocrine disorder that may cause polyneuropathy.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Proprioception | Pre-treatment, 2 weeks, 1 month
  Proprioception will be assessed using joint position sense. Joint position sense will be measured as the ability to actively replicate a joint position previously taught passively, referred to as Active Joint Position Sense (AJPS) (28). AJPS will be tested using a Continuous Passive Motion (CPM) device. The knee will be passively moved from 90° flexion toward extension at a slow pace. During this movement, the knee will be paused at 60°, 45°, and 30° flexion for 10 seconds each, and these angles will be taught to the participants. The knee will then be returned to 90° flexion, and the participants will be asked to actively replicate the taught angles.
  Participants will actively move their knees from the starting position to the taught angles of 60°, 45°, and 30° flexion to identify these positions. The actual taught angles and the angles determined by the participants will be recorded, and the differences between them will be calculated. Each angle will be tested in three trials, and

SECONDARY OUTCOMES:
The Nottingham Health Profile (NHP) | Pre-treatment, 2 weeks, 1 month
  The Nottingham Health Profile (NHP) will be used to assess quality of life. The NHP is a general quality of life questionnaire that measures perceived health problems and their impact on normal daily activities. The questionnaire consists of 38 items and evaluates six dimensions of health status: energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), and physical activity (8 items). Responses are given as "yes" or "no," and each section is scored on a scale from 0 to 100. A score of "0" indicates the best health status, while a score of "100" represents the worst health status.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Pre-treatment, 2 weeks, 1 month
  Pain, joint stiffness, and functional status will be assessed using the Western Ontario and McMaster Universities Arthritis Index (WOMAC). The WOMAC consists of 24 questions in total, divided into three subscales: pain (5 questions), joint stiffness (2 questions), and functional status (17 questions).
  Each question is scored on a scale from 1 to 5, with higher scores indicating poorer health and lower scores indicating better health.
Visual Analog Scale (VAS) | Pre-treatment, 2 weeks, 1 month
  Pain intensity will be assessed using the Visual Analog Scale (VAS) for evaluating current pain. Participants will be asked to rate their pain at rest, during movement, and at night. The scale ranges from 0 (no pain) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tuzun EH, Eker L, Aytar A, Daskapan A, Bayramoglu M. Acceptability, reliability, validity and responsiveness of the Turkish version of WOMAC osteoarthritis index. Osteoarthritis Cartilage. 2005 Jan;13(1):28-33. doi: 10.1016/j.joca.2004.10.010. PMID 15639634
- [Background] Myles PS, Troedel S, Boquest M, Reeves M. The pain visual analog scale: is it linear or nonlinear? Anesth Analg. 1999 Dec;89(6):1517-20. doi: 10.1097/00000539-199912000-00038. PMID 10589640
- [Background] Krcmery V. [Antibiotics and antimycotics in oncology]. Vnitr Lek. 1991 Jul-Aug;37(7-8):695-702. Slovak. PMID 1755212
- [Background] Pavlou M, Stefoski D. Development of somatizing responses in multiple sclerosis. Psychother Psychosom. 1983;39(4):236-43. doi: 10.1159/000287745. PMID 6635137
- [Background] Cortez VS, Moraes WA, Taba JV, Condi A, Suzuki MO, Nascimento FSD, Pipek LZ, Mattos VC, Torsani MB, Meyer A, Hsing WT, Iuamoto LR. Comparing dextrose prolotherapy with other substances in knee osteoarthritis pain relief: A systematic review. Clinics (Sao Paulo). 2022 May 17;77:100037. doi: 10.1016/j.clinsp.2022.100037. eCollection 2022. PMID 35594623
- [Background] Shanahan EM, Robinson L, Lyne S, Woodman R, Cai F, Dissanayake K, Paddick K, Cheung G, Voyvodic F. Genicular Nerve Block for Pain Management in Patients With Knee Osteoarthritis: A Randomized Placebo-Controlled Trial. Arthritis Rheumatol. 2023 Feb;75(2):201-209. doi: 10.1002/art.42384. Epub 2022 Nov 11. PMID 36369781
- [Background] Porzig H, Baer M, Chanton C. Properties of beta-adrenoceptor sites in metabolizing and nonmetabolizing rat reticulocytes and in resealed reticulocyte ghosts. Naunyn Schmiedebergs Arch Pharmacol. 1981;317(4):286-93. doi: 10.1007/BF00501308. No abstract available. PMID 6119626
- [Background] Liu SH, Dube CE, Eaton CB, Driban JB, McAlindon TE, Lapane KL. Longterm Effectiveness of Intraarticular Injections on Patient-reported Symptoms in Knee Osteoarthritis. J Rheumatol. 2018 Aug;45(9):1316-1324. doi: 10.3899/jrheum.171385. Epub 2018 Jun 15. PMID 29907665
- [Background] Mendes JG, Natour J, Nunes-Tamashiro JC, Toffolo SR, Rosenfeld A, Furtado RNV. Comparison between intra-articular Botulinum toxin type A, corticosteroid, and saline in knee osteoarthritis: a randomized controlled trial. Clin Rehabil. 2019 Jun;33(6):1015-1026. doi: 10.1177/0269215519827996. Epub 2019 Feb 19. PMID 30782000
- [Background] Steultjens MP, Dekker J, van Baar ME, Oostendorp RA, Bijlsma JW. Range of joint motion and disability in patients with osteoarthritis of the knee or hip. Rheumatology (Oxford). 2000 Sep;39(9):955-61. doi: 10.1093/rheumatology/39.9.955. PMID 10986299
- [Background] Cowan SM, Bennell KL, Hodges PW, Crossley KM, McConnell J. Delayed onset of electromyographic activity of vastus medialis obliquus relative to vastus lateralis in subjects with patellofemoral pain syndrome. Arch Phys Med Rehabil. 2001 Feb;82(2):183-9. doi: 10.1053/apmr.2001.19022. PMID 11239308
- [Background] Brandt KD, Heilman DK, Slemenda C, Katz BP, Mazzuca S, Braunstein EM, Byrd D. A comparison of lower extremity muscle strength, obesity, and depression scores in elderly subjects with knee pain with and without radiographic evidence of knee osteoarthritis. J Rheumatol. 2000 Aug;27(8):1937-46. PMID 10955336
- [Background] Felson DT, Lawrence RC, Hochberg MC, McAlindon T, Dieppe PA, Minor MA, Blair SN, Berman BM, Fries JF, Weinberger M, Lorig KR, Jacobs JJ, Goldberg V. Osteoarthritis: new insights. Part 2: treatment approaches. Ann Intern Med. 2000 Nov 7;133(9):726-37. doi: 10.7326/0003-4819-133-9-200011070-00015. PMID 11074906